CLINICAL TRIAL: NCT04007562
Title: Acute Rhabdomyolysis and Muscle Pain Associated With Mutations in the LPIN1 Gene - A Retrospective Study Describing the Safety and Efficacy of Hydroxychloroquine Sulfate Given on a Compassionate Basis to Patients Suffering From Lipin-1 Deficiency
Acronym: LIPIN-1-METAB
Status: Withdrawn | Type: Observational
Why Stopped: The study never started
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190368
Record Dates: First submitted 2019-05-29; First posted 2019-07-05 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2024-10

CONDITIONS: LIPIN1 Deficiency
Keywords: LIPIN1 deficiency; Acute episodes of rhabdomyolysis; Myoglobinuria; Hydroxychloroquine Sulfate; Orphan drug
MeSH Terms: conditions — Myoglobinuria | interventions — Hydroxychloroquine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lipin-1 deficiency: Patients suffering from Lipin-1 deficiency havebenefited from an off-label use treatment by Hydroxychloroquine Sulfate as part of their care for at least 6 months.
  Interventions: Drug: Hydroxychloroquine Sulfate

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate — The dosage and the route of administration of Hydroxychloroquine Sulfate was the same than in Lupus disease:
  Oral administration: administered in soluble form in patients under the age of 6 years old and administered in tablets in patients other the age of 6 years old with Lipin-1 deficiency.
  The soluble form was prepared at the Necker Hospital Pharmacy. Dose: 6.5 mg/kg/day (max 400 mg/day). The plasma concentration of the drug during follow-up was made, in order to follow a possible overdose.

SUMMARY:
Lipin-1 deficiencies are responsible for severe rhabdomyolysis and muscle pain in childhood. A specific treatment does not exist. Our research team (Pr de Lonlay, Pr Van-Endert, Marine Madrange and Perrine Renard) identified the mechanism of this disease and propose a treatment to decrease rhabdomyolysis outcome and muscle pain. Further to a CPP approval in 2015, several patients have been treated by Hydroxychloroquine Sulfate off label use on a compassionate basis.

The objective of this retrospective study is to describe the safety and efficacy of Hydroxychloroquine Sulfate given on a compassionate basis to patients suffering from Lipin-1 deficiency within a period between 6 and 36 months.

DETAILED DESCRIPTION:
The Lipin-1 deficiency is an inherited autosomal recessive disease caused by two mutations in the LPIN1 gene. Homozygous or compound heterozygous Lipin-1 deficiency causes recurrent acute episodes of rhabdomyolysis and myoglobinuria in children, associated with permanent muscle pain and weakness. The onset of the disease is usually early (before the age of 6 years old) and the disease is severe. The number of acute episodes' ranges from 1 to 10 per patient, mostly during the first 6 years of life (period where illness episodes are most frequent). Some patients die of myoglobinuric bouts, from cardiac arrhythmia, possibly due to hyperkalemia, with a heart probably more sensitive to hyperkaliemia. Mortality rate is around 10%, and is significantly higher when rhabdomyolysis is complicated by renal failure or by cardiac arrest with arrhythmia due to hyperkalemia. A specific treatment does not exist. Altogether these observations indicate that there is a crucial need to identify a treatment.

Our research team (Pr de Lonlay, Pr Van-Endert, Marine Madrange and Perrine Renard) identified the mechanism of this disease. The consequences on myoblasts of patients are TLR9 sequestration in late endosomes and mitophagy impairment, with consecutively mitochondrial DNA accumulation, TLR9 activation, inflammatory cytokines, calcium release and cell death in the presence of TLR9 ligands and a nutrient-poor environment.

Hydroxychloroquine Sulfate, thanks to an anti-TLR9 activity restores control cell phenotypes. In vivo and in vitro results are spectacular. This treatment seems to be able to both decrease the signaling cascade resulting from the activation of TLR9 and to correct the phenotype of patients suffering from the Lipin-1 deficiency.

Further to a CPP approval, several patients have been treated by Hydroxychloroquine Sulfate off label use on a compassionate basis. The objective of this retrospective study is to describe the safety and efficacy of Hydroxychloroquine Sulfate given on a compassionate basis to patients suffering from Lipin-1 deficiency within a period between 6 and 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 3 months
* Minors with Lipin-1 deficiency which were diagnosed with familiar context analysis followed by genetic diagnosis (two causal mutations on the LPIN1 gene) and treated by Hydroxychloroquine Sulfate off label use on a compassionate basis in the Metabolic Diseases Center of Necker Hospital
* Patients treated by Hydroxychloroquine Sulfate for at least 6 months

Exclusion Criteria:

- Opposition of parental authority holders

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population to be studied consists of 8 paediatric patients with Lipin-1 deficiency followed-up by the metabolic diseases center of Necker hospital and having been treated by Hydroxychloroquine sulfate for at least 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Creatine kinase dosage in plasma | 36 months
Inflammatory cytokines in plasma | 36 months
  Quantitative flow cytometry based mutliplex assays (flow cytometry-based systems (BD™ Cytometric Bead Array)).
Quantification of mitochondrial DNA in plasma | 36 months
  Quantitative PCR to detect mitochondrial DNA, 12s gene.

SECONDARY OUTCOMES:
Occurrence of intercurrent event | 36 months
  Clinical examination.
Occurrence of rash | 36 months
  Clinical examination.
Gowers sign appearance | 36 months
  Clinical examination.
Occurrence of shortness of breath | 36 months
  Clinical examination.
Occurrence of muscular fatigability | 36 months
  Clinical examination.
Treatment compliance | 36 months
  Patient interrogation.
Occurrence of adverse effect | 36 months
  Patient interrogation.
Dosing of Hydroxychloroquine Sulfate in plasma | 36 months
  Compliance.
Occurence of retinopathy. | 36 months
  Fundus eye and electroretinogram.
Quotation of the different muscles | 36 months
  Muscle testing by a physiotherapist.
6-min walking test | 36 months
Test of the number of steps during a 3-min walk | 36 months
Assessment of pain: VAS | 36 months
  Visual analogue scale (VAS) : scale from 1 to 10; compare from one examination to another for a patient (which is his own control).
Quality-of-life assessment: Pediatric Quality of Life InventoryTM (PedsQL) questionnaire | 36 months
  Pediatric Quality of Life InventoryTM (PedsQL) questionnaire adapted to age: child questionnaire and parent questionnaire. Questionnaire of 23 questions scored on 5 points, from 0 (never) to 4 (almost always). The scores are linearly transformed on a scale between 0 and 100, added together and divided by the number of items completed; high scores are associated with a better quality of life related to health.
Echocardiography | 36 months
  Measurement of the wall of the ventricles, ejection fraction.
Absence of cardiac arrhythmia | 36 months
  Electrocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Pascale de Lonlay, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Caroline Tuchmann-Durand, Pharm. D, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamel Y, Mauvais FX, Madrange M, Renard P, Lebreton C, Nemazanyy I, Pelle O, Goudin N, Tang X, Rodero MP, Tuchmann-Durand C, Nusbaum P, Brindley DN, van Endert P, de Lonlay P. Compromised mitochondrial quality control triggers lipin1-related rhabdomyolysis. Cell Rep Med. 2021 Aug 17;2(8):100370. doi: 10.1016/j.xcrm.2021.100370. eCollection 2021 Aug 17. PMID 34467247